CLINICAL TRIAL: NCT06172049
Title: Incidence of Colorectal Cancer in Southwest China: Based on SCC Database
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Clinical Professor, West China Hospital
Other Study IDs: CRC-2023
Record Dates: First submitted 2023-12-06; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRC cases
  Interventions: Other: treatment

INTERVENTIONS:
Other: treatment — the actual treatment CRC patients have reveived

SUMMARY:
To evaluate recent trends in CRC incidence, treatment, and survival in the Southwest China.

DETAILED DESCRIPTION:
The epidemiological feature of colorectal cancer (CRC) showed different trends among countries. Studying the epidemiological and management characteristics between China and the US has important implications for understanding the current status of cancer occurrence, treatment and survival. we established the Southwest China Colorectal (SCC) database, aiming to provide reference information on the diagnosis and management of CRC in China.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of colorectal cancer;
2. Received treatment in medical institutions;
3. Regular follow-up after the diagnosis.

Exclusion Criteria:

Patients who lost to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who were diagnosed with CRC were included
Sampling Method: Non-Probability Sample
Enrollment: 5838 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Survival | From inclusion until date of death from any cause, or untile the 2023-10-31
  Overall survival (OS) untile the end of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Wang, Study Chair — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No